CLINICAL TRIAL: NCT03930069
Title: Efficacy of Transcervical Vasopressin Injection VersusVaginal Misoprostol During Hysteroscopic Myomectomy in Reducing Operative Blood Loss and Operation Time: A Randomized Trial.
Brief Title: Vasopressin Injection Versus Misoprostol During Hysteroscopic Myomectomy In Reducing Blood Loss And Operation Time.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hossam mohamed, clinical investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hysterscopioc myomectomy
Record Dates: First submitted 2019-04-23; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Submucous Leiomyoma of Uterus
MeSH Terms: interventions — Misoprostol; Vasopressins

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- misoprostol group (Active Comparator): 20 cases received 400 microgram prostaglandin E1 analogue, misoprostol, (Misotac®, 200 microgram, by SIGMA pharmaceutical industries, Alexandria, Egypt), intra-vaginally, 2 hr before operation.
  Interventions: Drug: Misoprostol
- vasopressin group (Active Comparator): 20 patients who had hysteroscopic guided intralesional vasopressin injection before hysteroscopic myomectomy
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Misoprostol — prostaglandin E1 analogue vaginally inserted two hours before hystertsopic myomectomy to evaluate intraoperative blood loss and operative time needed for completion of myomectomy
  Other Names: Misotac
  Arms: misoprostol group
Drug: Vasopressin — one ampoule of vasopressin was diluted to 50 ml of normal saline, and 10 ml (4 units of vasopressin) was withdrawn in a syringe. Needle was inserted through the working channel of the hysteroscope until its tip was seen. The needle tip was pointed to the site of injection under hysteroscopic guidance during the whole injection technique. Aspiration was done first to avoid intravascular injection of vasopressin. The diluted solution was injected into the surface, especially to parts with dilated vasculature till they blanch.
  Arms: vasopressin group

SUMMARY:
A prospective randomized study designed to compare the efficacy of transcervical vasopressin injection versus vaginal misoprostol in reducing intra -operative blood loss during hysteroscopic mymectomy .

DETAILED DESCRIPTION:
This was a prospective, randomized, study on forty women with symptomatic submucous myoma presented mostly with bleeding and/or infertility scheduled for hysteroscopic myomectomy were randomized to groups (group A) 20 patients transcervical intramyoma vasopressin injection and (group B) 20patients with vaginal misoprostol is used .

ELIGIBILITY:
Inclusion Criteria:

* symptomatic women presented with bleeding or infertility and scheduled for hysterscopic myomectomy
* grade 0 and grade 1 submucous myomas
* less than 5 centimeters in diameter

Exclusion Criteria:

* Patients with grade 2 submucous myoma or more
* patients with submucous myomas larger than 5 cm in diameter
* postmenopausal women
* patients received GnRh analogue in last 6 months
* patients with anticoagulant therapy
* patients with endometrial premalignant or malignant pathologies
* patients with cardiovascular diseases, asthma or impaired kidney functions

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Yes: Eligibility is based on gender, As the subject of the study is hysterscopic myomectomy so the the clinical trial is based on female gender
Enrollment: 40 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
intraoperative bleeding | start with the first resectoscope myoma cut till withdrawal of hysterscope through the cervix at the end of the procedure
  subjective assessment of bleeding by the surgeon.
operative time | start with insertion of hysterscope through the cervix ends with withdrawal of hysterscopy through the cervix at the end of the procedure
  time needed for completion of myomectomy procedure
haemoglobin and hematocrit deficit | 24 hours before myomectomy and 24 hour after myomectomy
  haemoglobin and hematocrit values before and after myomectomy

SECONDARY OUTCOMES:
Degree of visual clarity | start with the first resectoscope myoma cut till the completion of myoma resection
  visual analogue scale straight horizontal line of fixed length, usually 100 mm and the ends are defined as the extreme limits of the parameter)
Fluid deficit | start with insertion of hysterscope through the cervix ends with withdrawal of hysterscopy through the cervix at the end pf the procedure
  calculation the fluid deficit between in flow volume and outflow volume
time need for cervical dilatation | start from grasping the cervix till insertion of hysterescope
  time needed to dilate the cervix to admit the operative hysterescope